CLINICAL TRIAL: NCT04479254
Title: The Impact of Indirect Calorimetry Guided Medical Feeding Protocol on Clinical Outcomes in Critically Ill Patients
Brief Title: The Impact of IC-Guided Feeding Protocol on Clinical Outcomes in Critically Ill Patients (The IC-Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Responsible Party: Principal Investigator, Mohd Basri Mat Nor, Associate.Professor, International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-504/14/11/2
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Critical Illness
Keywords: Indirect calorimetry, Energy expenditure, Critical illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indirect Calorimetry- Directed Nutrition (Experimental): Enteral Nutrition (EN) will be the preferred route of nutrition, and will be initiated within the first 24-48 hours of ICU admission. Caloric requirements will be measured by indirect calorimetry IC as soon as possible after recruitment and will be repeated in every 24 hrs. The amount of delivery is gradually increased to avoid the possibility of gastrointestinal intolerance. If EN fails to reach caloric goals or not feasible supplementary Parenteral nutrition(PN) will be initiated after 5-7days
  Interventions: Dietary Supplement: Enteral Nutrients ( Nutren Optimum, Nutren Diabetes, Novasource Renal ), Parenteral Nutrient ( Smofkabiven)
- Standard weight-based equation- Directed Nutrition (Active Comparator): Enteral Nutrition (EN) will be initiated within the first 24-48 hours of ICU. Admission. Enteral nutrient delivery is gradually increased to avoid the possibility of gastrointestinal intolerance so that a few days are required to achieve the caloric target. PN will be started after 5-7 days if EN is not feasible. Energy and protein goals will be calculated by the standard weight-based equation of 25 kcal/kg BW body weight and 1.2-2.5 g/kg body weight, respectively.
  Interventions: Dietary Supplement: Enteral Nutrients ( Nutren Optimum, Nutren Diabetes, Novasource Renal ), Parenteral Nutrient ( Smofkabiven)

INTERVENTIONS:
Dietary Supplement: Enteral Nutrients ( Nutren Optimum, Nutren Diabetes, Novasource Renal ), Parenteral Nutrient ( Smofkabiven) — Enteral nutrition feeding formula is used in powder form and will be reconstituted by attending nurses, Continuous feeding is commonly used which will be prescribed by the attending clinicians, Energy and protein intake from EN will be estimated by multiplying the volume of feed given to energy (kcal) and protein (g) in 1 ml of standard dilution, and for Standard PN product, energy and protein intake will also be calculated based on the volume infused.

SUMMARY:
Adequate nutritional support is an essential element for achieving favourable outcomes in critically ill patients. Therefore, an accurate determination of patients' energy needs is required to optimize nutritional support and reduce the harmful effects of under- and over-feeding. Currently, indirect calorimetry is considered as a gold standard for measuring energy expenditure during critical illness.

This randomized study aims to investigate the impact of indirect calorimetry guided nutrition therapy on clinical outcomes such as ICU. Mortality, hospital mortality, duration of mechanical ventilation, length of I.C.U./hospital stay and mascle wasting. The investigators hypothesis that nutrition therapy guided by IC will improve clinical outcomes in severely ill patients

DETAILED DESCRIPTION:
This is a single-blind randomized control study. Eligible participants are randomly assigned within 24 hrs of ICU. admission in two groups

* Intervention group: The calorie needs will be determined by indirect calorimetry.
* Control group: a routine standard weight-based equation (20-25kcal/kg ideal body weight/day) will be used to estimate the energy requirements of critically ill patients.

Daily energy and protein data will be recorded for a maximum of 12 evaluable days (nutritional days) or until death or discharge from ICU.while outcome data will be collected for a maximum of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged over 18 years old
* Critically ill patients with me ical ventilation
* Expected to have an ICU. stay of more than (3) days

Exclusion Criteria:

* Requirement for inspired oxygen content (FiO2) greater than 0.6
* Patients on high-frequency ventilation
* Patients with chest tubes that leak air/ Bronchopleural fistula
* Patients with incompetent tracheal cuff
* Patients inhaled nitric oxide therapy
* Patients receiving continuous renal replacement therapy (CRRT) during IC measurement
* Patients with pregnancy
* Patients with burn injury
* Patients infected with human immunodeficiency virus (HIV)
* Patients with severe liver disease (Child-Pugh score C)
* seizure activity
* patients suffering from significant head trauma (GCS <8)
* Patients with paraplegia and quadriplegia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-09-25 (Actual)

PRIMARY OUTCOMES:
ICU mortality | 28 Days
  Rate of mortality from all causes before or at day 28 in the ICU during the same ICU admission

SECONDARY OUTCOMES:
Length of ICU stay | 28 Days
  will be measured as the number of calendar days between admission and discharge from ICU.or until 28 days
Length of mechanical ventilation | 28Days
  will be measured as the calendar days between start and end of mechanical ventilation until 28 days
Length hospital stay | 28 Days
  will be calculated using the admission date and expiration or discharge date from hospital until 28 days
Hospital mortality | 28Days
  Rate of mortality from all causes (death in ICU or in ward) before or at day 28 during the same hospital admission.
Muscle wasting | First 10 days of ICU admission
  define as differences between the serial ultrasound measurement of quadriceps femoris muscle layer thickness (vastus intermedius and rectus femoris) over the first 10 days(on day 1,3,5,7 and 10 ) of ICU Admission.

CONTACTS AND LOCATIONS:
Overall Officials: DR. MOHD BASRI Mat Nor, M.Med (Anesthesiology), Principal Investigator — IIUM University
Locations (1):
- IIUM- Medical Center, Kuantan, Pahang, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer P, Anbar R, Cohen J, Shapiro H, Shalita-Chesner M, Lev S, Grozovski E, Theilla M, Frishman S, Madar Z. The tight calorie control study (TICACOS): a prospective, randomized, controlled pilot study of nutritional support in critically ill patients. Intensive Care Med. 2011 Apr;37(4):601-9. doi: 10.1007/s00134-011-2146-z. Epub 2011 Feb 22. PMID 21340655
- [Background] Allingstrup MJ, Kondrup J, Wiis J, Claudius C, Pedersen UG, Hein-Rasmussen R, Jensen TH, Lange T, Perner A. Early goal-directed nutrition in ICU patients (EAT-ICU): protocol for a randomised trial. Dan Med J. 2016 Sep;63(9):A5271. PMID 27585532